CLINICAL TRIAL: NCT02489461
Title: International, Multicenter, Randomized, Partially Blind Study to Evaluate Efficacy, Safety and Selection of the Optimal Dose for VM-1500 in Comparison to Efavirenz in Combination With Two NRTIs in Treatment-naïve, HIV-1 Infected Patients
Brief Title: Efficacy, Safety and Optimal Dose of VM-1500 in Comparison to Efavirenz Added to Standard-of-care Antiretroviral Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIV-VM1500-04
Record Dates: First submitted 2015-06-18; First posted 2015-07-03 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: HIV-1-infection
Keywords: HIV
MeSH Terms: interventions — elsulfavirine; efavirenz; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VM-1500 20 mg + ART (Experimental): VM-1500 - 20 mg (Stage I), then optimal dose (Stage II and Open-Label Stage), ART
  Interventions: Drug: VM-1500; Drug: Antiretroviral therapy (ART)
- VM-1500 40 mg + ART (Experimental): VM-1500 - 40 mg (Stage I), then optimal dose (Stage II and Open-Label Stage), ART
  Interventions: Drug: VM-1500; Drug: Antiretroviral therapy (ART)
- Efavirenz 600 mg + ART (Active Comparator): Efavirenz 600 mg (Stage I and Stage II), ART
  Interventions: Drug: Efavirenz; Drug: Antiretroviral therapy (ART)

INTERVENTIONS:
Drug: VM-1500 — VM-1500 up to 96 weeks
  Other Names: Elsulfavirine; Elpida®
  Arms: VM-1500 20 mg + ART; VM-1500 40 mg + ART
Drug: Efavirenz — Efavirenz up to 48 weeks
  Other Names: Stocrin®
  Arms: Efavirenz 600 mg + ART
Drug: Antiretroviral therapy (ART) — Antiretroviral therapy up to 96 weeks
  Other Names: standard antiretroviral therapy of two NNRTIs

SUMMARY:
The study is conducted in two stages and open-label stage of the study.

At the first stage of the study, the main purpose was to choose the optimal dose of VM-1500 (20 mg or 40 mg per day) in addition to standard-of-care basic antiretroviral therapy consisting of two NRTIs, in terms of reduction of viral load at Week 12 (<400 copies/ml) in treatment-naïve HIV-1-infected patients.

At the second stage of the study, the main purpose was to evaluate efficacy of VM- 1500 (in the optimal dose selected at the first stage of the study) in comparison to Efavirenz added to standard-of-care antiretroviral therapy of two NRTIs, in terms of reduction of viral load at Week 24 to the undetectable level (<50 copies/ml) in treatment-naïve HIV-1 infected patients.

Open-label stage of the study continued evaluation of viral load and immunological and safety parameters in HIV-1 patients receiving VM-1500 up to Week 96 and additional PK up to Week 100.

DETAILED DESCRIPTION:
This project is an international, multicenter, randomized, partially blind clinical study to evaluate efficacy and safety of two different doses of VM-1500 in comparison with Efavirenz added to standard antiretroviral therapy including two NRTIs in treatment-naïve HIV-1-infected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Patient Information and Informed Consent Form.
2. Males and females, age ≥ 18 years.
3. HIV-1 infection, confirmed serologically in IFA or immunoblot analysis (or documented HIV-1 infection).
4. Clinically stable HIV infection (clinical stages 1 or 2 according to the WHO classification).
5. Indications (in the Investigator's opinion) for ART, according to the WHO Summary Guideline for use of antiretroviral drugs in HIV prevention and treatment (2013).
6. HIV-1 RNA plasma level ≥ 5 000 copies/ml at screening.
7. СD4+ Т-cells number > 200 cells/mm3 at screening.
8. Laboratory parameters as follows:

White blood cells ≥ 2900/mm3 (2,9 x 109 cells/l) Absolute neutrophils ≥ 1500/mm3 (1,5 x 109 cells/l) Platelets ≥ 100000/mm3 (100 x 109 cells/l) Hemoglobin ≥ 9.0 g/dl Total bilirubin ≤ 1.5 x ULN AST and ALT≤ 2.5 x ULN Renal function GFR > 60 ml/min

Exclusion Criteria:

1. Primary HIV-1 resistance to ART. Viral resistance mutations are defined as any basic mutations of resistance to NNRTIs, according to the updated list of VIH-1 resistance mutations (International AIDS society, 2013), associated with drug resistance in any genotype.
2. History of antiretroviral therapy (ART), including for the prevention of vertical transmission of HIV.
3. Acute hepatitis or hepatic cirrhosis of any etiology; anti-HCV antibodies or HBsAg at screening.
4. Signs of acute infection or positive test result for syphilis, hepatitis A, Toxoplasma gondii, cytomegalovirus, gonorrhea, Chlamydia trachomatis during 30 days before screening.
5. Opportunistic infections of the Category C (Centers of Disease Control (CDC), 2008), excluding Kaposi's sarcoma not requiring systemic therapy.
6. History of tuberculosis of any localization, or tuberculosis at screening, according to x-ray examination.
7. History of malignant tumors (except basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ, eliminated and cured ≥ 5 years ago).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Reduction of HIV-1 RNA level in blood plasma <400 copies/ml | 12 weeks
  Comparison of the percentage of patients with reduced viral load to < 400 copies/ml at Week 12 in VM-1500 20 mg, VM-1500 40 mg and Efavirenz treatment groups

SECONDARY OUTCOMES:
Reduction of HIV-1 RNA level in blood plasma <50 copies/ml | 24 weeks
  Comparison of the percentage of patients with reduced viral load to an undetectable level (< 50 copies/ml) at Week 24 in VM-1500 group with the selected dose and Efavirenz group.
Reduction of HIV-1 RNA level in blood plasma <50 copies/ml | 48 weeks
  Comparison of the percentage of patients with reduced viral load to an undetectable level (< 50 copies/ml) at Week 48 in VM-1500 group with the selected dose and Efavirenz group.
Change in the absolute CD4+ lymphocytes count | 48 weeks
  Change in the absolute CD4+ lymphocytes count from Baseline to Week 48 in VM-1500 group with the selected dose and Efavirenz group.
Change in the absolute CD8+ lymphocytes count | 48 weeks
  Change in the absolute CD8+ lymphocytes count from Baseline to Week 48 in VM-1500 group with the selected dose and Efavirenz group.
The percent of patients with study therapy-resistant HIV-1 development | 48 weeks
  The proportion of patients who develop study therapy-resistant HIV-1 from Baseline to Week 48 in VM-1500 group with the selected dose and Efavirenz group.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Y Tyrnova, Study Chair — Viriom,LLC
Locations (13):
- Russia (13):
  - Kaluga regional center for AIDS prevention, Kaluga, Kaluga Oblast
  - Lipetsk regional center for AIDS prevention, Lipetsk, Lipetsk Oblast
  - Perm Regional center for AIDS prevention, Perm, Perm Krai
  - Ryazan Regional Clinical Dermatovenerologic Dispensary, Ryazan, Ryazan Oblast
  - City center for AIDS prevention, Tolyatti, Samara Oblast
  - Republican hospital for AIDS prevention, Kazan', Tatarstan Republic
  - Udmurtia Republican hospital for AIDS prevention, Izhevsk, Udmurtia Republic
  - Volgograd regional center for AIDS prevention, Volgograd, Volgograd Oblast
  - Central Scientific Research Institute of Epidemiology, Moscow
  - Moscow Infectional Clinical Hospital #2, Moscow
  - Moscow Prevention AIDS Center, Moscow
  - St.Petersburg city center for AIDS prevention, Saint Petersburg
  - Clinical infectious diseases hospital n.a. S.P. Botkin", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No